CLINICAL TRIAL: NCT01750905
Title: A Phase I, Randomized, Double-blind, Placebo-controlled, Crossover Study Evaluating The Safety, Hemodynamic And Neurohumoral Effects of a Novel Chimeric Peptide, CD-NP, in Patients With Left Ventricular Assist
Brief Title: Safety Study of Chimeric Natriuretic Peptide(CD-NP) in Stable LVAD Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John A. Schirger, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 12-001869
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Left Ventricular Insufficiency
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CD-NP (Active Comparator): CD-NP 5 ug/kg subcutaneous injection (SQ)
  Interventions: Drug: CD-NP
- Placebo (Placebo Comparator): Placebo: Vehicle (D5W) SQ
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CD-NP — CD-NP 5 ug/kg subcutaneous injection (SQ)
  Arms: CD-NP
Drug: Placebo — Vehicle (D5W) SQ
  Arms: Placebo

SUMMARY:
The most promising chimeric natriuretic peptide designed and studied by our group has been CD-NP which has anti-fibrotic and cardioprotective properties in vivo, vitro and in normal volunteers and human heart failure patients. Since left ventricular assist device (LVAD) can not reverse remodeling of the heart whereas it can improve hemodynamics, CD-NP may be novel anti-fibrotic and anti-remodeling drug as co-therapy during LVAD support.

DETAILED DESCRIPTION:
This study is a double blind, placebo-controlled phase I trial of the safety and neurohumoral activity of CD-NP, in the treatment of heart failure with LVAD support. Subjects more than 3 months after LVAD implantation will be screened at outpatient clinic visit appointments lists and interested qualified subjects will be either confronted at a visit or sent a letter in the mail to be consented and offered participation in this trial. Once consent has been obtained, baseline values will be established at day 1 and subjects will be given subcutaneous injection of placebo or CD-NP and stay overnight on two different visits in the Clinical Research Unit (CRU). Participant's will receive both placebo and the CD-NP during the study, one per visit. A final follow-up visit for clinical assessment will be conducted over the phone at the end of the study.

Potential subjects who present to Mayo Clinic, Rochester, Minnesota for follow up clinical visit after LVAD implantation will be identified by the study coordinator. A $300 remuneration per subject will be involved to compensate for the inconvenience to the subject. A $500 reimbursement of gas mileage will be provided for those who travel.

ELIGIBILITY:
Inclusion Criteria

* Male and non-pregnant/post-menopausal female, ages 18-90, in end-stage Heart Failure (HF) with LVAD support who are stable in the healed stage after at least 3 months from the LVAD implant (Destination therapy only) (the post-menopausal state is defined as the absence of menses for ≥ 1 year and serum follicle-stimulating hormone ≥ 20 IU/L; sterilization in the female is defined as bilateral tubal occlusion for ≥ 6 months, bilateral oophorectomy, or complete hysterectomy)
* Be willing to provide informed consent.

Exclusion Criteria

* Known allergy or other adverse reactions to exogenous natriuretic peptides (CD-NP or its components, nesiritide, other natriuretic peptides, or related compounds).
* Women who are pregnant, or breast-feeding.
* Having received nesiritide within 7 days prior to prior to entry into the study.
* Having received any investigational drug or device within 30 days prior to entry into the study.
* Clinically unstable patients (e.g. mean blood pressure < 70 mmHg, ongoing requirement for vasopressors, or mechanical ventilation).
* Recent hospitalization for decompensated HF or recent defibrillation for cardiac resuscitation within 30 days prior to randomization.
* Patients with guarded prognosis who are unlikely to derive meaningful benefit from CD-NP.
* Use of sulfonamides, non-steroidal anti-inflammatory drugs, probenecid, or other drugs that are known to alter renal function within one week of the first dose of CD-NP or placebo.
* Presence of cardiac lesions or comorbidities that may contraindicate the use of natriuretic peptides, such as clinically significant cardiac valvular stenosis, hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, primary pulmonary hypertension, or uncorrected congenital heart disease that contraindicates the use of vasodilators.
* Symptomatic carotid artery disease, known critical carotid stenosis, or stroke within the past 3 months
* Clinically significant renal artery stenosis
* Baseline hemoglobin < 9.0 g/dl.
* Serum sodium < 130 mEq/L, potassium < 3.6 milliequivalents per Liter (mEq/L), or magnesium < 1.5 mEq/L.
* Elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) at least 5 times the upper limit of normal or bilirubin at least 5 times the upper limit of normal
* Creatinine clearance (CrCl) < 30 ml.min-1.1.73m-2, as calculated by Cockcroft-Gault formula(35) and adjusted for body surface area within 3 months or at screening, or requirement for dialysis.
* History of alcohol or drug abuse within the past 6 months.
* Inability to communicate effectively with study personnel.
* BMI >40

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-04; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Hypotension | approx day 9

SECONDARY OUTCOMES:
Mean plasma Cyclic guanosine monophosphate (cGMP) level | Approx day 9
Mean aldosterone level | approx 9 days

CONTACTS AND LOCATIONS:
Overall Officials: John Schirger, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No